CLINICAL TRIAL: NCT06909539
Title: Using a Perineometer Device With Gamification to Improve Symptom Outcomes in Pediatric Pelvic Floor Dysfunction
Brief Title: HOme PElvic Floor Improvement Trainer Trial
Acronym: HoPE FIT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24-1026
Record Dates: First submitted 2025-03-27; First posted 2025-04-03 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Pelvic Pain; Pelvic Floor Dysfunction; Voiding Dysfunction
Keywords: voiding dysfunction; pelvic floor dysfunction; pelvic pain; perineometer; gamification
MeSH Terms: conditions — Pelvic Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Voiding Dysfunction (Experimental): Patients with voiding dysfunction only and no pelvic pain symptoms will use the home pelvic floor trainer daily for 2 months.
  Interventions: Device: Home Pelvic Floor Trainer
- Pelvic pain (Experimental): Patients with pelvic pain with or without voiding dysfunction symptoms will use the home pelvic floor trainer daily for 2 months.
  Interventions: Device: Home Pelvic Floor Trainer

INTERVENTIONS:
Device: Home Pelvic Floor Trainer — The intervention utilizes a perineometer device with biofeedback features.
  This device employs external electrodes to measure pelvic floor muscle strength. It then provides real-time feedback through a smartphone application during exercise sessions. The application uses gamification to engage users and track progress. Patients can choose between two games: a bird game or a space-themed game. In the bird game, patients activate their pelvic floor muscles to make the bird fly upward. In the space game, pelvic floor contractions fire a laser or activate a shield. A visual bar displays the strength of pelvic floor contractions. Games are designed to be played for 5 minutes daily, 7 days a week, with increasing difficulty as the user progresses through levels.

SUMMARY:
This study will gauge the efficacy of a home biofeedback treatment device for pelvic floor dysfunction/voiding dysfunction and pelvic pain. Investigators will test the utility of this device as a treatment alternative and/or temporary treatment for a patient's symptoms prior to or perhaps in lieu of their physical therapy appointment.

DETAILED DESCRIPTION:
This study aims to determine if a special device can help children with pelvic floor problems. The pelvic floor issues under investigation include difficulty controlling urination and ongoing pain in the lower belly. The study will explore whether the device helps children gain better control over urination.

It will also investigate if the device contributes to the reduction of pelvic pain experienced by children. Furthermore, the study will analyze if the device leads to improvement in how the body functions during urination. The consistency with which children use the device and adhere to instructions will be monitored. Finally, the study includes an assessment of whether children find the device acceptable for use.

ELIGIBILITY:
Inclusion Criteria:

* Dysfunctional voiding symptoms without chronic pelvic pain.
* Chronic pelvic pain with or without dysfunctional voiding symptoms.
* Daytime enuresis, nocturnal enuresis, frequency, urgency, dysuria
* 8 years - 18 years, no one under 8 and no one over 18.

Exclusion Criteria:

- Has seen a physical therapist for traditional physical therapy of the pelvic floor due to urinary symptoms or chronic pelvic pain within the last 12 months.

Note: This would include patients who begin physical therapy for their pelvic floor outside of the study while enrolled in the study.

-All patients with the following conditions: severe developmental delay such as CP or wheelchair bound, cannot eat by mouth, mechanical ventilation dependence, etc.

* Nonverbal or unable to effectively communicate needs and preferences.
* Within the voiding dysfunction group, a diagnosis of a congenital GU anomaly (bladder exstrophy, cloacal anomaly, spina bifida, etc.)
* No initial medication usage will be excluded; however, if the patient begins a new medication or treatment regimen during the study, the patient will be excluded.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Dysfunctional Voiding symptom scale (30 point scale) | 0 weeks baseline, 4 weeks, and 8 weeks patients will take the DVSS survey
  this survey will be given to all participants and is the primary outcome of the DV group. This will be attained at the initial urology consult visit, 4-week, and 8-week visits. The DVSS is a 30 point scale with higher scores representing more severe voiding dysfunction symptoms. Males with score greater than 9 points are considered to have voiding dysfunction, and females with score greater than 6 are considered to have voiding dysfunction.
McGill Pain Scale (Short Form- points scale) | 0 weeks baseline, 4 weeks, and 8 weeks patients will take the McGill pain Scale Short Form survey
  this survey will be given to all participants and is the primary outcome of the Pelvic Pain group. This will be attained at the initial urology consult visit, 4-week, and 8-week visits. total of 22 items with 0-10 numerical response options, 0 being no pain and the higher score representing more pain)

SECONDARY OUTCOMES:
Post-Void Residual Volume (mL) | 0 weeks baseline, 8 weeks in-person visits investigators will attain PVR
  PVR volume > 10% normal will be considered elevated PVR. This will be attained from all participants at an initial baseline urology visit as part of standard of care, and the 8-week in-person visit.
Uroflowmetry | Investigators will attain uroflowmetry at the same time as the PVR measurement, at initial baseline (0 weeks) and last (8 weeks) in-person visits.
  Uroflowmetry parameters will be assessed at the initial and 8-week visits. These parameters include:
  A normal, bell-shaped curve.
  A tower flow curve, suggesting detrusor overactivity.
  A staccato flow curve, suggesting external sphincter activity.
  An intermittent or interrupted flow curve, suggesting underactive detrusor or dysfunctional voiding.
  A plateau shape curve, suggesting bladder outlet obstruction

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Harris, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Skardoon GR, Khera AJ, Emmanuel AV, Burgell RE. Review article: dyssynergic defaecation and biofeedback therapy in the pathophysiology and management of functional constipation. Aliment Pharmacol Ther. 2017 Aug;46(4):410-423. doi: 10.1111/apt.14174. Epub 2017 Jun 29. PMID 28660663
- [Background] Vasconcelos M, Lima E, Caiafa L, Noronha A, Cangussu R, Gomes S, Freire R, Filgueiras MT, Araujo J, Magnus G, Cunha C, Colozimo E. Voiding dysfunction in children. Pelvic-floor exercises or biofeedback therapy: a randomized study. Pediatr Nephrol. 2006 Dec;21(12):1858-64. doi: 10.1007/s00467-006-0277-1. Epub 2006 Sep 12. PMID 16967285
- [Background] Wagner B, Steiner M, Huber DFX, Crevenna R. The effect of biofeedback interventions on pain, overall symptoms, quality of life and physiological parameters in patients with pelvic pain : A systematic review. Wien Klin Wochenschr. 2022 Jan;134(Suppl 1):11-48. doi: 10.1007/s00508-021-01827-w. Epub 2021 Mar 22. PMID 33751183
- [Background] Taylor AS, Cabo JJ, Lauderdale C, Maskan N, Thomas JC, Tanaka ST, Pope JC, Adams MC, Brock JW, Shannon CN, Clayton DB. Pelvic floor biofeedback therapy in children: Assessment of symptom scores in responders and non-responders. Neurourol Urodyn. 2019 Jan;38(1):254-260. doi: 10.1002/nau.23842. Epub 2018 Oct 23. PMID 30350888